CLINICAL TRIAL: NCT01011907
Title: Characterizing Alpha5 Nicotinic Receptors in Alcohol and Nicotine Dependence
Brief Title: A Pilot Clinical Trial of Varenicline as a Treatment for Alcohol Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: EGCRC0109; RC2AA019429 (NIH)
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Results first posted 2013-02-25 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Substance Dependence
MeSH Terms: conditions — Substance-Related Disorders | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- varenicline (Experimental): Drug: varenicline (Chantix) 12 weeks of oral tablet treatment in an escalating dosing regimen (0.5 mg 1x daily, days 1-3; 0.5mg 2x daily, days 4-7, 1.0 mg 2x daily, days 8-84).
  Interventions: Drug: varenicline
- placebo (Placebo Comparator): Drug: placebo for varenicline 12 weeks of oral tablet treatment in an escalating dosing regimen (1 - 2x daily).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — 12 weeks of oral tablet treatment in an escalating dosing regimen (0.5 mg 1x daily, days 1-3; 0.5mg 2x daily, days 4-7, 1.0 mg 2x daily, days 8-84).
  Other Names: Chantix
  Arms: varenicline
Drug: placebo — 12 weeks of oral tablet treatment in an escalating dosing regimen (1 - 2x daily).
  Arms: placebo

SUMMARY:
Purpose: This is an outpatient, randomized, double-blinded, placebo-controlled study in which either varenicline (twice daily) or placebo will be administered over a 12 week study period to examine genetic influences on treatment response to varenicline for reduction of hazardous drinking.

DETAILED DESCRIPTION:
Hazardous alcohol use and alcohol use disorders (AUDs) are an area of large unmet medical needs. Although there has been some progress with pharmacotherapy for alcohol-dependent individuals, a critical need for the development of novel and additional therapeutic approaches remains. Pharmacotherapy development for AUDs as a therapeutic area has had several recent advancements, where clinically as well as commercially successful additions to available treatment options are available and several more are expected in the near future. Based on recent preclinical work, we believe that varenicline has potential to become one of the first among those newly evolving treatments.

In this study, participants with nicotine dependence will receive standard varenicline or placebo treatment over the recommended course of 12 weeks. Since our research question addresses whether alcohol drinking also diminishes with varenicline treatment, we will not ask participants to alter alcohol use; we will simply follow their use over time. Study visits will take place at the Ernest Gallo Clinic and Research Center. The procedures to be completed include vital signs, blood samples at screening and end of study, urine toxicology screening and the completion of standard questionnaires. No special facilities are required for these procedures. Group therapy (which is not a research procedure, but part of standard nicotine dependence treatment) will take place at the Gallo Center.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 75 years.
* Currently seeking treatment for nicotine dependence (smoke at least 10 cigarettes daily) and found to have problem drinking, alcohol abuse or alcohol dependence (non-physiological) as determined by amount of alcohol consumed weekly (Average weekly alcohol consumption (last 30 days), >7 standard drinks (for women) or >14 standard drinks (for men), clinical interview, and AUDIT score > 8.
* Generally healthy, without serious or unstable medical/mental illness(es).
* Smokers only will be included (degree of nicotine dependence will be assessed and included in analysis).
* Able to give voluntary, written, informed consent

Exclusion Criteria:

* More than 30 days of abstinence from alcohol in the prior 90 days.
* History of major alcohol-related complications within the preceding 2 years (liver failure/cirrhosis, pancreatitis, esophageal varices, liver function tests > 3 X ULN).
* Intolerance to the study medication.
* Current psychiatric disorder(s) requiring clinical treatment.
* Any recent history (i.e. within the preceding 5 years) of suicide attempt or current suicidal ideation.
* Use of illicit or non-prescribed psychotropic drug use (opiates, benzodiazepines, cocaine, PCP, methamphetamine, cocaine, or marijuana more than twice a week).
* A history of complicated alcohol or other drug withdrawal syndrome(s), e.g.: delirium tremens or seizures.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Fields, MD PhD, Principal Investigator — UCSF: Ernest Gallo CLinic and Research Center; Jennifer Mitchell, PhD, Study Director — UCSF: Ernest Gallo Clinic and Research Center
Locations (1):
- UCSF: Ernest Gallo Clinic and Research Center, Emeryville, California, United States

REFERENCES:
- [Result] Mitchell JM, Teague CH, Kayser AS, Bartlett SE, Fields HL. Varenicline decreases alcohol consumption in heavy-drinking smokers. Psychopharmacology (Berl). 2012 Oct;223(3):299-306. doi: 10.1007/s00213-012-2717-x. Epub 2012 May 1. PMID 22547331

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 99 subjects were consented of which 64 successfully completed the screening process were randomized to treatment. Results are posted for the 35 subjects who completed the study.
Groups:
- Placebo: Drug: placebo for varenicline 12 weeks of oral tablet treatment in an escalating dosing regimen (1 - 2x daily).
  placebo : 12 weeks of oral tablet treatment in an escalating dosing regimen (1 - 2x daily).
- Varenicline: Drug: varenicline (Chantix) 12 weeks of oral tablet treatment in an escalating dosing regimen (0.5 mg 1x daily, days 1-3; 0.5mg 2x daily, days 4-7, 1.0 mg 2x daily, days 8-84).
  varenicline : 12 weeks of oral tablet treatment in an escalating dosing regimen (0.5 mg 1x daily, days 1-3; 0.5mg 2x daily, days 4-7, 1.0 mg 2x daily, days 8-84).
Period: Overall Study
Arm/Group | Placebo | Varenicline
Started | 31 | 33
Completed | 17 | 18
Not Completed | 14 | 15
Not completed — Withdrawal by Subject | 13 | 11
Not completed — Adverse Event | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Varenicline | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Cigarettes Smoked Between the Varenicline and Placebo Groups for Completers Through Week 12.
Time Frame: Weeks 1-12
Measure: Mean (Standard Error); unit: cigarettes
Arm/Group | Placebo | Varenicline
Number analyzed (Participants) | 17 | 18
cigarettes | 788.94 (96.27) | 403.24 (102.42)

2. Secondary Outcome: Average Number of Alcoholic Drinks Consumed Between the Varenicline and Placebo Groups for Completers of the Study Through Week 12.
Time Frame: Weeks 1-12
Measure: Mean (Standard Error); unit: drinks
Arm/Group | Placebo | Varenicline
Number analyzed (Participants) | 17 | 17
drinks | 277.5 (41.9) | 177.04 (28.86)

3. Secondary Outcome: Alcohol Craving as Measured by the Obsessive Compulsive Drinking Scale (OCDS) Between Varenicline and Placebo Groups for Completers of the Study.
Description: Higher scores on the OCDS indicate increased craving. OCDS possible score range = 0 - 40. Difference in average OCDS scores from week 1 to week 12 were reported for the varenicline and placebo groups in subjects that completed the study.
Time Frame: Week 1 to Week 12
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Varenicline
Number analyzed (Participants) | 17 | 18
Scores on a scale | -3.07 (0.389) | -4.36 (0.205)

ADVERSE EVENTS:
Arm/Group | Placebo | Varenicline
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | Varenicline (N=33)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No